CLINICAL TRIAL: NCT05494268
Title: Effects of Preoperative Oral Carbohydrate Loading on Maternal Thiol-disulfide Homeostasis
Status: Completed | Type: Observational
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ozlem Dulger, Assist Prof, Karamanoğlu Mehmetbey University
Other Study IDs: KaramanogluMehmeybeyU
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy Related; Cesarean Delivery Affecting Fetus; Fetus Fetus
MeSH Terms: conditions — Fetus-in-Fetu | interventions — Carbohydrates

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental ( Carb Group): Preoperative education will be provided by researchers to the patients on the ward before fluid intake. Solid food will be forbidden starting at 20:00 p.m, and drinking will be forbidden after 22:00 p.m the day before surgery. The Carb Group will consume carbohdrate fluid and Non-carb Group will consume equal amount of water at night and two hours before the surgery.
  Interventions: Drug: Carbohydrate
- Standart Care (Non-carb Group): Preoperative education will be provided by researchers to the patients on the ward before fluid intake. Solid food will be forbidden starting at 20:00 p.m, and drinking will be forbidden after 22:00 p.m the day before surgery. The Carb Group will consume carbohdrate fluid and Non-carb Group will consume equal amount of water at night and two hours before the surgery.

INTERVENTIONS:
Drug: Carbohydrate — Preoperative Carbohydrate Loading Drink
  Groups: Experimental ( Carb Group)

SUMMARY:
The primary aim of this randomised control trial is to assess the impact of pre-operative carbohydrate loading on thiol disulfide homeostasis when compared to standard care in elective cesarean section. Half of the participants will receive pre-operative carbohydrates and the other half will receive standard care.

DETAILED DESCRIPTION:
The concept of enhanced recovery after surgery (ERAS) has been gradually extended from surgery to the field of obstetrics. Carbohydrate loading before the surgery in obstetric patients reduce the incidence of nausea and vomiting and reduce insulin resistance. Although these effects of the preoperative carbohydrate loading has been studied, the thiol disulfide homeostasis effects after carbohydrate loading has not been investigated yet. Thiol-disulfide homeostasis (TDH) plays a critical role in the mechanisms of antioxidant defense, detoxification, apoptosis, regulation of enzyme activities, transcription, and cellular signal transduction. Since the newborns are very susceptible to harmfull effects of reactive oxygen species, the effect of carbohydrate loading on the reactive oxygen species gain importance.

All mothers undergoing a planned caesarean section in the Karaman Training and Research Hospital will be invited to participate. Mothers will be divided into two groups. One group will receive standard care and the other group will receive a carbohydrate drink in addition to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancies,
* Planned elective ceserean sections,
* Under spinal anesthesia,
* Pregnants who can read and write Turkish.

Exclusion Criteria:

* Preterm pregnants,
* Pregnants with reflux,
* obesity,
* hiatus hernia,
* ileus,
* enteral nutrition,
* alcohol or substance abuse,
* prolonged delivery,
* systemic chronic diseases,
* malignancy,
* GDM,eclampsia,preeclampsia,
* fetal anomaliy,
* prolonged delivery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only pregnant patients will be studies.
Study Population: The term pregnant patients admitted to Karaman Training and Research Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-05 (Actual)

PRIMARY OUTCOMES:
The comparison of the changes in thiol disulfide values between the groups | From beginning to two hours after the surgery
  The native thiol, total thiol, disulfide, native thiol/total thiol ratio, disulfide/native thiol ratio, and disulfide/total thiol ratio will be determined.

SECONDARY OUTCOMES:
Incidence of intraoperative hypotension | From beginning to the end of the surgery
  Hypotension is defined as a decrease in the mean arterial pressure by ˃20% of the baseline value.
Total ephedrine usage | From beginning to the end of the surgery
  At hypotensive episodes, 5 mg ephedrine will be used intravenously.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Dulger, Assist Prof, Principal Investigator — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All the results of the study will be shared on request.